CLINICAL TRIAL: NCT04305639
Title: The Reliability and Validity of Turkish Version of ''The Dyspnea-ALS-Scale (DALS-15)"
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: IstanbulMU4
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Dyspnea
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Dyspnea-ALS-Scale (DALS-15) is a uni-dimensional scale to measure dyspnea in patients with Amyotrophic Lateral Sclerosis. It can be easily and rapidly applied. The aim of this study is to investigate reliability and validity of Turkish version of the DALS-15.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or above
* Dyspnea on exertion, dyspnea at rest, or orthopnea without evidence of pulmonary or cardiac causes of dyspnea

Exclusion Criteria:

* Severe cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with Amyothrophic Lateral Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
The Dyspnea-ALS-Scale (DALS-15) | 10 minutes
  The scale is used to measure dyspnea in ALS patients

SECONDARY OUTCOMES:
Modified Borg Scale | 10 minutes
  A 10 point Modified Borg Scale is used to assess dyspnea in supine and standing positions.
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) | 15 minutes
  It is used to assess functional stats in ALS patients. This study particularly focus on pulmonary functions and dyspnea subscale of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: ESMA NUR KOLBAŞI, MSc, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No